CLINICAL TRIAL: NCT06114277
Title: The Relationship Between Intraoperative ETCO2 Levels and Postoperative Pain and Nausea-Vomiting in Laparoscopic Robotic Prostatectomy Patients
Brief Title: The Relationship Between Intraoperative ETCO2 Levels and Postoperative Pain and Nausea-Vomiting
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Özgüner, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: AnkaraEtlikYusufOzguner005
Record Dates: First submitted 2023-10-29; First posted 2023-11-02 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative; Nausea, Postoperative; Vomiting, Postoperative
Keywords: End-tidal carbon dioxide; Laparoscopic Robotic Prostatectomy
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with low ETCO2 levels: Intraoperative ETCO2 values between 26 and 35 in laparoscopic robotic prostatectomy patients were included in this group.
  Interventions: Other: ETCO2 levels
- Patients with high ETCO2 levels: Intraoperative ETCO2 values between 36 and 45 in laparoscopic robotic prostatectomy patients were included in this group.
  Interventions: Other: Patients with high ETCO2 levels

INTERVENTIONS:
Other: ETCO2 levels — Intraoperative ETCO2 values between 26 and 35 in laparoscopic robotic prostatectomy patients were included in group 1.
  Other Names: Patients with low ETCO2 levels
  Groups: Patients with low ETCO2 levels
Other: Patients with high ETCO2 levels — Intraoperative ETCO2 values between 36 and 45 in laparoscopic robotic prostatectomy patients were included in group 2.
  Groups: Patients with high ETCO2 levels

SUMMARY:
The aim of our study is to investigate the relationship between intraoperative ETCO2 levels and postoperative nausea-vomiting and pain scores in patients undergoing robotic laparoscopic radical prostatectomy. The investigators will monitor patients' 24-hour postoperative pain, nausea-vomiting and the consumption of additional analgesic and antiemetic medications.

DETAILED DESCRIPTION:
Robotic surgery provides several advantages in the field of surgery, including a three-dimensional view of the surgical site, the elimination of surgeon hand tremors, and enhanced precision in movements. Additionally, it offers benefits such as reduced intraoperative bleeding, faster return to daily functions for patients, and decreased hospitalization duration. Consequently, the use of robots in various surgical procedures has become widespread in contemporary medical practice.

Robot-assisted laparoscopic radical prostatectomy is a surgical technique performed in a head-down Trendelenburg position with intraperitoneal insufflation of carbon dioxide (CO2). This positioning and pneumoperitoneum lead to an increase in intraabdominal pressure, as well as elevated intracranial and intraocular pressures.

End-tidal carbon dioxide (ETCO2) levels can vary during laparoscopic surgery. An increase in ETCO2 levels has been reported to cause an elevation in intracranial pressure, leading to an increased incidence of postoperative nausea and vomiting. Some studies in the literature have investigated the relationship between ETCO2 values and the incidence of postoperative nausea and vomiting in patients. Furthermore, it is believed that hypercarbia (elevated carbon dioxide levels) may have an impact on postoperative pain.

The aim of our study is to investigate the relationship between intraoperative ETCO2 levels and postoperative nausea, vomiting, and pain scores in patients undergoing robotic laparoscopic radical prostatectomy. The investigators will monitor patients' 24-hour postoperative pain, nausea, vomiting, and the consumption of additional analgesic and antiemetic medications.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between the ages of 18 and 80.
2. Patients with American Society of Anesthesiologists (ASA) scores I, II, or III.
3. Patients who have undergone robotic laparoscopic prostatectomy in the operating room.

Exclusion Criteria:

1. Patients under 18 years old or over 80 years old.
2. Patients with American Society of Anesthesiologists (ASA) scores IV and above.
3. Patients who refuse to participate in the study.
4. Patients undergoing emergency surgery.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Robotic prostate surgery is a procedure performed on male patients.
Study Population: The aim of our study is to investigate the relationship between intraoperative ETCO2 levels and postoperative nausea, vomiting, and pain scores in patients undergoing robotic laparoscopic radical prostatectomy. We will monitor patients' 24-hour postoperative pain, nausea, vomiting, and the consumption of additional analgesic and antiemetic medications.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting (PONV) Score | 0-2-4-8-12-24 hours postoperatively
  Postoperative nausea and vomiting recording in patients.
  * 0=no PONV: patient reports no nausea and has had no emesis episodes;
  * 1=mild PONV: patient reports nausea but declines antiemetic treatment;
  * 2=moderate PONV: patient reports nausea and accepts antiemetic treatment; and
  * 3=severe PONV: nausea with any emesis episode (retching or vomiting). Higher scores indicate severe postoperative nausea and vomitting.

SECONDARY OUTCOMES:
Pain on the Numeric Rating Scale (NRS) | 0-2-4-8-12-24 hours postoperatively
  Participants recorded pain rated on the numeric rating scale (NRS) at 6 time points. NRS range was from 0-10 with 0 being no pain and 10 the worst pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Ozguner, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Varlık Mahallesi, Halil Sezai Erkut Caddesi Yenimahalle, Turkey (Türkiye)

REFERENCES:
- [Result] Aceto P, Beretta L, Cariello C, Claroni C, Esposito C, Forastiere EM, Guarracino F, Perucca R, Romagnoli S, Sollazzi L, Cela V, Ercoli A, Scambia G, Vizza E, Ludovico GM, Sacco E, Vespasiani G, Scudeller L, Corcione A; Societa Italiana di Anestesia Analgesia Rianimazione e Terapia Intensiva (SIAARTI), Societa Italiana di Ginecologia e Ostetricia (SIGO), and Societa Italiana di Urologia (SIU). Joint consensus on anesthesia in urologic and gynecologic robotic surgery: specific issues in management from a task force of the SIAARTI, SIGO, and SIU. Minerva Anestesiol. 2019 Aug;85(8):871-885. doi: 10.23736/S0375-9393.19.13360-3. Epub 2019 Mar 29. PMID 30938121
- [Result] Besir A, Tugcugil E. Comparison of different end-tidal carbon dioxide levels in preventing postoperative nausea and vomiting in gynaecological patients undergoing laparoscopic surgery. J Obstet Gynaecol. 2021 Jul;41(5):755-762. doi: 10.1080/01443615.2020.1789961. Epub 2020 Oct 12. PMID 33045886
- [Result] Son JS, Oh JY, Ko S. Effects of hypercapnia on postoperative nausea and vomiting after laparoscopic surgery: a double-blind randomized controlled study. Surg Endosc. 2017 Nov;31(11):4576-4582. doi: 10.1007/s00464-017-5519-8. Epub 2017 Apr 7. PMID 28389799